CLINICAL TRIAL: NCT03058770
Title: Study of the Effect of a Sensorimotor Retraining Program in Chronic Stroke
Brief Title: Sensorimotor Retraining in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, M. Arantzazu Ruescas Nicolau, Doctor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H14831 09435066
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: chronic stroke, sensorimotor retraining
MeSH Terms: conditions — Stroke | interventions — Relaxation Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sensorimotor retraining program (Experimental): Fifteen 40-minute sensorimotor retraining sessions will be provided over a 5-week period.
  Interventions: Other: Sensorimotor retraining
- Relaxation technique (Active Comparator): Subjects will perform fifteen 40-minute relaxation sessions over a 5-week period.
  Interventions: Other: Relaxation technique

INTERVENTIONS:
Other: Sensorimotor retraining — Subjects will receive education regarding sensation and sensory retraining; practice in detection and localization of touch and in discrimination of hardness, texture and temperature in sitting and standing with vision obscured; proprioception training; and practice of these sensations in functional activities.
  Arms: sensorimotor retraining program
Other: Relaxation technique — Subjects will perform guided relaxation by using the Jacobson technique.
  Arms: Relaxation technique

SUMMARY:
A prospective, randomized double-blind clinical trial will be conducted to determine the effect of a sensorimotor retraining program on the sensory and functional recovery of the paretic lower limb of subjects with chronic sequelae from stroke.

DETAILED DESCRIPTION:
Somatosensory deficits are a common symptom after stroke, affecting a high percentage of survivors (50-80%). These impairments have a long-term influence on somatosensory capacity, motor ability and functional performance. Although several authors have studied the effect of sensorimotor retraining on recovery of the paretic upper limb, a few have investigated its effect on the paretic lower limb. Furthermore, most of them have done so in the acute and subacute phases after stroke. Thus, in this field there is a lack of studies of high methodological quality that provide effective physiotherapeutic interventions, especially in chronic stroke.

On the other hand, the importance of motor recovery of the paretic lower limb in order to achieve a better balance, gait and independence in the activities of daily living is well established. In this regard, sensory loss in the feet may difficult effective motor function recovery due to its impacts upon ambulatory activity. After stroke, sensory dysfunction in the lower limb has been related to reductions in static and dynamic balance as well as in gait speed and symmetry. Therefore, successful recovery of sensory function after stroke may allow for the appropriate integration of sensory inputs in order to maintain balance and adapt to changing environmental demands during gait.

Since the current evidence indicates that there may be recovery of sensory loss during the chronic phase of stroke, the present study aims to evaluate the effect of a sensorimotor retraining program on sensory and functional recovery of the paretic lower limb in chronic stroke. The investigators hypothesized that stroke survivors receiving the somatosensory training program would demonstrate significantly greater improvement in sensation, static and dynamic balance and gait pattern in comparison with the control intervention.

To cope with the objective of the study, a prospective randomized double-blind clinical trial will be conducted. By means of advertisements in supporting groups, rehabilitation facilities and the external consultations of various hospitals, subjects who meet the inclusion criteria will be recruited. After screening and giving signed consent, participants will be randomly allocated to the intervention group or the control group. In addition to the usual physical activity, participants will complete fifteen 40-minute sessions of sensorimotor retraining (intervention group) or of Jacobson relaxation (control group) over a 5-week period. Participants will be assessed prior to treatment and on completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemiplegia or hemiparesis from a first ever stroke (onset > 6 months prior to study enrolment)
* No severe cognitive deficit (Mini-Mental State Examination score ≥ 22)
* Subjective reports of sensory loss
* Triceps surae muscles scoring ≤ 2 on the Modified Ashworth Scale
* Able to walk for at least 10 meters indoor over ground without assistance

Exclusion Criteria:

* Ataxia
* Co-existing sensory deficits from peripheral neuropathies (i.e. diabetes mellitus)
* Lower extremity claudication
* Pain > 3/10 on a visual analogue scale
* Prior lower extremity surgical history
* Blindness, visual impairments and other pathologic condition that influence posture and balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Light touch | 6 weeks
  Von Frey monofilaments

SECONDARY OUTCOMES:
Static balance | 6 weeks
  Stabilometric parameters (Romberg test (eyes open and close) and the limits of stability test in 8 directions) registered on the NedSVE/IBVv4 force plate system
Plantar pressure distribution | 6 weeks
  Percentage of weight supported under each foot during upright position and the symmetry ratio between feet assesed by using computerized baropodometric analysis.
Gait | 6 week
  Biomechanical analysis of the ground reaction forces, gait speed and single leg supporting time registered on the NedSVE/IBVv4 force plate system.

CONTACTS AND LOCATIONS:
Overall Officials: M. Arántzazu Ruescas-Nicolau, PhD, Principal Investigator — University of Valencia; M.Luz Sanchez-Sanchez, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain